CLINICAL TRIAL: NCT03836963
Title: Cognitive Rehabilitation for Veterans With Parkinson's Disease
Brief Title: Cognitive Rehab for Parkinson's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N3015-P; RX003015 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2019-01-28; First posted 2019-02-11 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: Parkinson's disease; cognition; cognitive training; prospective memory; executive function
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: randomized control trial. three arms to the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cognitive and memory strategy training (Experimental): The cognitive training will include 4 sessions/week for 8 weeks. Each session will take 30min. Total hours of training is 16 hours. For memory strategy training, strategies will be performed daily; this will take only a few minutes a day to accomplish.
  Interventions: Behavioral: cognitive training; Behavioral: memory strategy training
- cognitive and memory strategy control training (Active Comparator): The cognitive training will include 4 sessions/week for 8 weeks. Each session will take 30min. Total hours of training is 16 hours. For the active control of memory strategy training, strategies will be performed daily; this will take only a few minutes a day to accomplish.
  Interventions: Behavioral: cognitive training; Behavioral: memory strategy training
- active control for cognitive and memory strategy training (Active Comparator): The cognitive training will include 4 sessions/week for 8 weeks. Each session will take 30min. Total hours of training is 16 hours. For the active control of memory strategy training, strategies will be performed daily; this will take only a few minutes a day to accomplish.
  Interventions: Behavioral: active control cognitive training; Behavioral: memory strategy training

INTERVENTIONS:
Behavioral: cognitive training — Cognitive training consists of a set of computerize games played on an iPad at home. Training will include 4 sessions/week for 8 weeks. Each session will take 30min. Total hours of training is 16 hours.
  Arms: cognitive and memory strategy control training; cognitive and memory strategy training
Behavioral: active control cognitive training — The active control consists of a set of computerized games played on an iPad. Training will include 4 sessions/week for 8 weeks. Each session will take 30min. Total hours of training is 16 hours.
  Arms: active control for cognitive and memory strategy training
Behavioral: memory strategy training — the participant's prospective memory strategies will be developed with researchers. Participants will be engage in the strategies daily; this will take only a few minutes a day to accomplish.
  Arms: cognitive and memory strategy training
Behavioral: memory strategy training — the participant's prospective memory strategies will be developed with researchers. Participants will be engage in the strategies daily; this will take only a few minutes a day to accomplish.
  Arms: active control for cognitive and memory strategy training; cognitive and memory strategy control training

SUMMARY:
This study will examine the feasibility of an at-home cognitive training program that incorporates both memory training and online computerized cognitive training (CCT) software. Data will also be collected to determine if this program improves thinking and memory as well as everyday function. The hypothesis is that memory and cognitive training combined , compared to memory training alone or will lead to greater improvements in cognitive performance and daily function.

DETAILED DESCRIPTION:
The objective of this study is to examine feasibility of an at-home cognitive rehabilitation program that incorporates both prospective implementation intentions strategies (PRIIS) and an existing web-based executive function (EF) computerized cognitive training (CCT) software for Veterans with Parkinson's disease (PD) and to collect pilot data to determine the impact of this program on cognition and everyday function. The central hypothesis is that CCT+PRIIS, compared to CCT alone and an active control group, will lead to greater improvements in cognitive performance and daily function. This innovative study uses a set of on-line training games that target aspects of EF susceptible in PD and trains the transfer of cognitive benefits to everyday function, using PRIIS, for Veterans with PD and mild cognitive impairment in executive function. Additionally, training is conducted at home allowing for convenience and flexibility for participants.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who seek services at Hines VA Hospital
* Diagnosis of PD as determined by the UK Parkinson's Disease Society Brain Bank Diagnostic Criteria
* Meet criteria for having mild cognitive impairment
* Receiving stable (i.e., no changes in medication and medication dose) medication and who are expected to remain on stable medication for the duration of the RCT
* 50 years or older
* Speak and read English

Exclusion Criteria:

* Dementia
* Failure to demonstrate decision making capacity
* Cholinesterase inhibitor medication
* History of deep brain stimulation surgery
* Severe depression
* Severe anxiety
* Severe apathy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L. Kletzel, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw and/or normalized data will be made available in the form of Excel files.
Time Frame: Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available.
Access Criteria: These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive and Memory Strategy Training | Cognitive and Memory Strategy Control Training | Active Control for Cognitive and Memory Strategy Training
Started | 2 | 1 | 3
Completed | 1 | 1 | 2
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive and Memory Strategy Training | Cognitive and Memory Strategy Control Training | Active Control for Cognitive and Memory Strategy Training | Total
Number analyzed (Participants) | 2 | 1 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [59 to 76] | 74 [74 to 74] | 74 [73 to 76] | 72 [59 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 1 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 1 | 3 | 5
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3 | 6
Montreal Cognitive Assessment [Mean (Full Range); unit: units on a scale] — Total MoCA score can range from 0-31. Higher scores indicate better global cognitive performance. Scores between 21-25 screen for mild cognitive impairment.
  units on a scale | 25.5 [25 to 26] | 21 [21 to 21] | 21 [21 to 22] | 22 [21 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Change in NIH Sponsored Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (NIH-EXAMINER) Executive Composite Score
Description: The NIH-EXAMINER has an established 3-factor model defined by (1) cognitive control, (2) working memory (3) fluency. A confirmatory factor analysis indicates these 3-factors load on to 1-factor: executive composite score. Seven tests in the NIH-EXAMINER is used to compute the composite score. -3 and +3 are the minimum and maximum values. Higher scores indicated better performance.
Time Frame: week 0 (before intervention begins), 8 weeks
Population: Only 4 participants completed the intervention and were assessed at endpoint. NIH-EXAMINER is a computerized assessment and must be completed in person. Due to the COVID-19 pandemic, not all assessments could be done in person. Only 2 participants who completed the intervention were able to be assessed with the NIH-EXAMINER in person. No participants randomized to the the Cognitive and Memory Strategy Control Training completed an endpoint NIH-EXAMINER assessment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive and Memory Strategy Training | Active Control for Cognitive and Memory Strategy Training
Number analyzed (Participants) | 1 | 1
units on a scale | 0.34 (0) | -.42 (0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cognitive and Memory Strategy Training | Cognitive and Memory Strategy Control Training | Active Control for Cognitive and Memory Strategy Training
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03836963/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT03836963/ICF_000.pdf